CLINICAL TRIAL: NCT03885726
Title: Assessing Clinical Effect of HVNI on Patient Ambulation in Acute Care Scenarios: a Feasibility Study
Brief Title: HVNI Ambulation Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: Knox Community Hospital (Other); Riverside Medical Center (Other); Midwest Chest Consultants (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RP-VTPF2018001Sci
Record Dates: First submitted 2019-02-25; First posted 2019-03-22 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Insufficiency; Dyspnea
MeSH Terms: conditions — Respiratory Insufficiency; Dyspnea | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment as Usual (Active Comparator)
  Interventions: Device: Treatment as Usual
- High Velocity Nasal Insufflation (Experimental)
  Interventions: Device: Precision Flow Plus

INTERVENTIONS:
Device: Precision Flow Plus — High velocity nasal insufflation
  Arms: High Velocity Nasal Insufflation
Device: Treatment as Usual — Conventional therapy per institution
  Arms: Treatment as Usual

SUMMARY:
The pilot/feasibility study evaluates the ability of High Velocity Nasal Insufflation (HVNI) therapy to facilitate ambulation and mobilization in patients experiencing shortness of breath, as compared to simple oxygen therapy.

DETAILED DESCRIPTION:
The hypothesis is that HVNI therapy, when implemented in conjunction to ambulatory practices, will be more effective than TAU to improve patient mobility by reducing the patient's perceived dyspnea and exertion via maintaining oxygenation (reduced desaturation) and supporting ventilation (reduced work of breathing [WOB]). The primary endpoint is exercise performance, defined as the distance and duration of patient ambulation.

To provide a sample data set, The investigators will enroll up to 32 subjects to complete this feasibility assessment, with a calculated sample size of N=26 plus a 20% failure rate. This will provide sufficient initial data to inform the appropriate sample size of a follow-on randomized study.

This will be a feasibility study, performed as a prospective, crossover controlled trial to evaluate the potential patient improvement during ambulation while on HVNI relative to TAU. Patients who fit the criteria for inclusion will perform ambulation for each study arm: the control arm (TAU) followed by the test arm (HVNI). Control group will receive the site TAU (not HVNI), and the test group will receive HVNI therapy. In both cases the clinical management will otherwise remain unchanged based on the site SOC practices. The patient FiO2 and flow values will be recorded while on any supplemental oxygen. Subjects will wear appropriate gear and, when applicable, have mobile carts to provide supplemental oxygen therapy (e.g. HVNI VTU) during ambulation. If they meet criteria for intubation or are deemed to need intubation by the critical care team, they will undergo prompt intubation and be managed according to standard practice. After each of the study arms, the clinicians will complete perception score assessments.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Demonstrated respiratory distress upon mild to moderate exertion (e.g. dyspnea upon standing, walking, etc.)
* Candidate for clinical ambulation/mobilization

Exclusion Criteria:

* Hypoxemia at resting baseline: unable to maintain SpO2≥88% with supplemental oxygen
* Inability to provide informed consent
* Pregnancy
* Known contraindication to perform ambulation, per site SOC practices
* Inadequate respiratory drive or any known contraindications to HVNI
* Inability to use nasal cannula and HVNI therapy
* Agitation or uncooperativeness
* Determined by the attending clinician to be sufficiently unstable or unsuitable for this feasibility study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shailesh Patel, MD, Principal Investigator — Knox Community Hospital; Thomas M Siler, MD, Principal Investigator — Midwest Chest Consultants; Paragkumar Amin, MD, Principal Investigator — Riverside Medical Center
Locations (3):
- United States (3):
  - Midwest Chest Consultants, Saint Charles, Missouri
  - Knox Community Hospital, Mount Vernon, Ohio
  - Riverside Regional Medical Center, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place in both an inpatient hospital setting and an outpatient medical clinic setting.
Pre-assignment Details: Of the N=32 enrolled patients, only N=28 completed both study arms. An additional N=3 patients were excluded from study analysis, making the total number of patient data analyzed post-hoc N=25.
Groups:
- All Study Participants: Crossover study design with the first intervention as "Treatment as Usual - 6 minute walk test" (TAU), followed by an adequate recovery period. The second intervention was "High Velocity Nasal Insufflation - 6 minute walk test" (HVNI). The patient population for both treatment arms was represented by both inpatients and outpatients.
Period: Overall Study
Arm/Group | All Study Participants
Started | 32
Completed | 28
Not Completed | 4
Not completed — Staffing issues/lost interest | 1
Not completed — Early discharge from hospital | 3

BASELINE CHARACTERISTICS:
Population: N=32 patients were enrolled in the study; of those, N=28 completed both study arms. A total of N=25 were analyzed post-hoc.
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 68.3]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Out of the N=28 patients who completed both arms of the study, N=3 were excluded post-hoc, making the total analysis population N=25.
  Participants
    Female | 12
    Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: N=32 patients were enrolled in the study; of those, N=28 completed both study arms. A total of N=25 were analyzed post-hoc.
  participants
    United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Exercise Performance- Distance
Description: Defined as the distance of patient ambulation
Time Frame: Through study completion, an average of 1 day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: meters
Groups:
- Treatment as Usual (Inpatient); Treatment as Usual (Outpatient): Treatment as Usual: Conventional therapy per institution
- High Velocity Nasal Insufflation (Inpatient); High Velocity Nasal Insufflation (Outpatient): Precision Flow Plus: High Velocity Nasal Insufflation
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
meters | 78.8 [63 to 144.1] | 88.6 [75.3 to 172.6] | 182.9 [134.1 to 453.4] | 165.2 [136.9 to 455.2]

2. Primary Outcome: Exercise Performance- Duration
Description: Defined as the duration of patient ambulation
Time Frame: Through study completion, an average of 1 day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
seconds | 211.5 [139.5 to 376.5] | 229.5 [164.3 to 387] | 307 [192.5 to 452.5] | 250 [180 to 537]

3. Secondary Outcome: Patient Recovery Interval
Description: Defined as recovery time (return time to baseline rated perceived dyspnea).
Time Frame: Through study completion, an average of 1 day
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
seconds | 283.5 [232 to 462.3] | 191.5 [172 to 395.5] | 239 [143 to 330] | 245 [135.5 to 359.5]

4. Secondary Outcome: Patient Vital Signs - Blood Pressure
Description: Patient blood pressure (systolic) measured in mmHg
Time Frame: Through study completion, an average of 1 day
Population: Of N=32 enrolled patients, N=28 completed both study arms, and N=3 were excluded post-hoc, making the analyzed population N=25.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
mmHg | 125.5 [119.8 to 152.5] | 137 [114.8 to 141.5] | 129 [120 to 132] | 113 [110 to 120]

5. Secondary Outcome: Patient Vital Signs-- Heart Rate [HR]
Description: Heart rate in bpm
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: beats per minute (bpm)
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
beats per minute (bpm) | 101 [88.3 to 108.3] | 94 [89.8 to 103.5] | 81 [72 to 89] | 79 [75 to 82]

6. Secondary Outcome: Patient Vital Signs-- Respiratory Rate [RR]
Description: Respiratory rate in breaths per minute
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: breaths per minute (brpm)
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
breaths per minute (brpm) | 20 [17.5 to 20] | 18 [17.5 to 20] | 20 [18 to 20] | 20 [18 to 20]

7. Secondary Outcome: Patient Vital Signs-- Arterial Oxygen Saturation
Description: SpO2 measured as percentage of oxygen saturation (%).
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation (%)
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
percentage of oxygen saturation (%) | 95 [93 to 97.3] | 95 [93 to 98] | 95 [94 to 95] | 95 [93 to 97]

8. Secondary Outcome: Patient Vital Signs-- Rated Perceived Exertion (RPE)
Description: Patient's subjective assessment of their exertion, rated as a modified Borg score on a scale from 0 to 10 . Higher scores indicate a worse outcome.
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
score on a scale | 1.5 [0 to 3] | 0.5 [0 to 1.25] | 0 [0 to 0.5] | 0.5 [0 to 0.5]

9. Secondary Outcome: Patient Vital Signs-- Rated Perceived Dyspnea (RPD)
Description: Patient's subjective assessment of their dyspnea, rated as a modified Borg score on a scale from 0 to 10. Higher scores indicate a worse outcome.
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
score on a scale | 0.5 [0 to 2] | 0.75 [0 to 1] | 0 [0 to 0.5] | 0 [0 to 0]

10. Secondary Outcome: Clinician Perception Score- Patient Response to Therapy
Description: Clinician's subjective assessment of the patient's clinical response to the therapy, rated as units on a visual analog scale from 0 to 100. A lower score indicates a better outcome.
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
units on a scale | 44.5 [3.38 to 69.5] | 8.25 [1.13 to 61.5] | 9 [3 to 49.5] | 37.5 [15 to 58.5]

11. Secondary Outcome: Clinician Perception Score- Patient Tolerance and Comfort
Description: Clinician's subjective assessment of the patient's comfort on and tolerance of the therapy, rated as units on a visual analog scale from 0 to 100. Lower values indicate a better outcome.
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
units on a scale | 33.8 [1.75 to 69.3] | 4 [1.25 to 17.1] | 1 [0 to 20.5] | 19 [8.5 to 82]

12. Secondary Outcome: Clinician Perception Score- Frequency of Technical/Clinical Difficulties
Description: Clinician's subjective assessment of the frequency of technical or clinical issues during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
units on a scale | 1.5 [1 to 4.5] | 1.5 [0.5 to 6.38] | 1 [0 to 2.5] | 3 [0.5 to 17.5]

13. Secondary Outcome: Clinician Perception Score- Simplicity of Set-up and Use
Description: Clinician's subjective assessment of the the simplicity of setting up and using the equipment, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 1 day
Population: Of the N=32 patients enrolled in the study, N=28 completed all study arms. An additional N=3 were excluded from post-hoc analysis, making the final analysis N=25.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
units on a scale | 1 [0.25 to 2.25] | 1.5 [0 to 2.5] | 1 [0.5 to 2.75] | 2 [0.75 to 3]

14. Secondary Outcome: Clinician Perception Score- Support/Adjustment Required
Description: Clinician's subjective assessment of the amount of support and adjustment required from the clinician during the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 13 | 16 | 9 | 9
units on a scale | 2 [0.25 to 11.3] | 2 [0.5 to 20.3] | 18.5 [1 to 33.8] | 18.5 [0.5 to 48.3]

15. Secondary Outcome: Patient Vital Signs - Blood Pressure
Description: Patient blood pressure (diastolic) measured in mmHg
Time Frame: Through study completion, an average of 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Treatment as Usual (Inpatient) | High Velocity Nasal Insufflation (Inpatient) | Treatment as Usual (Outpatient) | High Velocity Nasal Insufflation (Outpatient)
Number analyzed (Participants) | 16 | 16 | 9 | 9
mmHg | 2 [0.25 to 11.3] | 2 [0.5 to 20.3] | 18.5 [1 to 33.8] | 18.5 [0.5 to 48.3]

ADVERSE EVENTS:
Time Frame: 8 hours
Arm/Group | Treatment as Usual | High Velocity Nasal Insufflation
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03885726/Prot_SAP_000.pdf